CLINICAL TRIAL: NCT00928408
Title: PRIMARA: A Prospective Descriptive Observational Study to Review Mimpara (Cinacalcet) Use in Patients With Primary Hyperparathyroidism in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20070363; PRIMARA
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2015-09

CONDITIONS: Hyperparathyroidism, Primary
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Cinacalcet

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cinacalcet
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet

SUMMARY:
This is a multicentre, descriptive observational study of adult patients with primary HPT receiving cinacalcet in clinical practice in a number of countries in Europe. Patients will be enrolled within 1 month of initiating cinacalcet treatment, and data will be collected prospectively for up to 1 year from initiation. Data will continue to be collected from patients discontinuing cinacalcet before the end of this period.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age at the time of first administration of cinacalcet
* patients with primary HPT who have initiated cinacalcet within 1 month before enrolment in the study
* provision of informed consent (if required)

Exclusion Criteria:

* previous use of cinacalcet (other than within 1 month before enrolment)
* diagnosed secondary HPT
* other known aetiology of hypercalcaemia (eg, sarcoidosis, tuberculosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with primary HPT receiving cinacalcet in clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Langdahl BL, Ralston SH. Diagnosis and management of primary hyperparathyroidism in Europe. QJM. 2012 Jun;105(6):519-25. doi: 10.1093/qjmed/hcr225. Epub 2012 May 7. PMID 22566664
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cinacalcet
Started | 305 (Number Enrolled)
Full Analysis Set | 303 (All enrolled participants who fulfilled the study inclusion/exclusion criteria)
Completed | 282
Not Completed | 23
Not completed — Other | 2
Not completed — Withdrawal by Subject | 4
Not completed — Death | 5
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241
  Male | 62
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0
  Black or African American | 0
  Unknown or Not Reported | 104
  White or Caucasion | 199

OUTCOME MEASURES:

1. Primary Outcome: Cinacalcet Dose
Description: Cinacalcet dose at initiation of treatment
Time Frame: Initiation of treatment
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
mg/day | 43.9 (0.9) [42.1 to 45.7]

2. Primary Outcome: Cinacalcet Dose
Description: Cinacalcet dose at Month 3
Time Frame: Month 3
Population: Full Analysis Set - Participants with Observed Data
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | Cinacalcet
Number analyzed (Participants) | 255
mg/day | 48.7 (0.9) [44.9 to 52.5]

3. Primary Outcome: Cinacalcet Dose
Description: Cinacalcet dose at Month 6
Time Frame: Month 6
Population: Full Analysis Set - Participants with Observed Data
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | Cinacalcet
Number analyzed (Participants) | 233
mg/day | 48.9 (0.9) [44.9 to 52.8]

4. Primary Outcome: Cinacalcet Dose
Description: Cinacalcet dose at Month 12
Time Frame: Month 12
Population: Full Analysis Set - Participants with Observed Data
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | Cinacalcet
Number analyzed (Participants) | 219
mg/day | 51.3 (0.9) [47.0 to 55.5]

5. Primary Outcome: Cinacalcet Dose
Description: Cinacalcet dose at end of treatment (last dose received)
Time Frame: Up to Month 12
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
mg/day | 53.1 (0.9) [49.2 to 57.0]

6. Primary Outcome: Cinacalcet Dosing Frequency
Description: Cinacalcet dosing frequency at initiation of treatment
Time Frame: Initiation of treatment
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
Participants
  Once a day | 169 (0.9) [49.2 to 57.0]
  Twice a day | 134

7. Primary Outcome: Cinacalcet Dosing Frequency
Description: Cinacalcet dosing frequency at Month 3
Time Frame: Month 3
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 255
Participants
  Once a day | 133 (0.9) [49.2 to 57.0]
  Twice a day | 107
  Three times a day | 4
  Four times a day | 1
  Dose withheld | 6
  Other | 4

8. Primary Outcome: Cinacalcet Dosing Frequency
Description: Cinacalcet dosing frequency at Month 6
Time Frame: Month 6
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 233
Participants
  Once a day | 128 (0.9) [49.2 to 57.0]
  Twice a day | 94
  Three times a day | 4
  Dose withheld | 3
  Other | 4

9. Primary Outcome: Cinacalcet Dosing Frequency
Description: Cinacalcet dosing frequency at Month 12
Time Frame: Month 12
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 219
Participants
  Once a day | 121 (0.9) [49.2 to 57.0]
  Twice a day | 88
  Three times a day | 6
  Other | 4

10. Primary Outcome: Cinacalcet Dosing Frequency
Description: Cinacalcet dosing frequency at end of treatment
Time Frame: Up to Month 12
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
Participants
  Once a day | 168 (0.9) [49.2 to 57.0]
  Twice a day | 118
  Three times a day | 10
  Four times a day | 3
  Other | 4

11. Primary Outcome: Occurrence of a Change in Cinacalcet Dose or Frequency During the First 3 Months After Initiation
Time Frame: Initiation to Month 3
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
Participants
  Yes | 100 (0.9) [49.2 to 57.0]
  No | 203

12. Primary Outcome: Occurrence of a Change in Cinacalcet Dose or Frequency >3 to 6 Months After Initiation
Time Frame: >3 to 6 months after initiation
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 255
Participants
  Yes | 45 (0.9) [49.2 to 57.0]
  No | 210

13. Primary Outcome: Occurrence of a Change in Cinacalcet Dose or Frequency >6 Months After Initiation
Time Frame: >6 months after initiation
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 233
Participants
  Yes | 51 (0.9) [49.2 to 57.0]
  No | 182

14. Primary Outcome: Duration of Exposure to Cinacalcet
Description: Time from first dose to last non-zero dose on study
Time Frame: 12 months
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
Days | 366 (7.3) [232 to 366]

15. Primary Outcome: Achievement of a Reduction From Baseline of Albumin-corrected Serum Calcium ≥ 0.25 mmol/L (1 mg/dL) at Month 3
Description: Baseline is pre-cinacalcet.
Time Frame: Month 3
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 180
Participants
  Yes | 101 (0.9) [49.2 to 57.0]
  No | 79

16. Primary Outcome: Achievement of a Reduction From Baseline of Albumin-corrected Serum Calcium ≥ 0.25 mmol/L (1 mg/dL) at Month 6
Description: Baseline is pre-cinacalcet.
Time Frame: Month 6
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 152
Participants
  Yes | 95 (0.9) [49.2 to 57.0]
  No | 57

17. Primary Outcome: Achievement of a Reduction From Baseline of Albumin-corrected Serum Calcium ≥ 0.25 mmol/L (1 mg/dL) at Month 12
Description: Baseline is pre-cinacalcet.
Time Frame: Month 12
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 117
Participants
  Yes | 70 (0.9) [49.2 to 57.0]
  No | 47

18. Primary Outcome: Incidence of an Albumin-corrected Serum Calcium Concentration ≤ 2.6 mmol/L (10.3 mg/dL) at Month 3
Time Frame: Month 3
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 220
Participants
  Yes | 138 (0.9) [49.2 to 57.0]
  No | 82

19. Primary Outcome: Incidence of an Albumin-corrected Serum Calcium Concentration ≤ 2.6 mmol/L (10.3 mg/dL) at Month 6
Time Frame: Month 6
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 193
Participants
  Yes | 134 (0.9) [49.2 to 57.0]
  No | 59

20. Primary Outcome: Incidence of an Albumin-corrected Serum Calcium Concentration ≤ 2.6 mmol/L (10.3 mg/dL) at Month 12
Time Frame: Month 12
Population: Full Analysis Set - Participants with Observed Data
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 148
Participants
  Yes | 105 (0.9) [49.2 to 57.0]
  No | 43

21. Primary Outcome: Change From Baseline to Month 3 in Albumin-corrected Serum Calcium
Time Frame: Baseline to Month 3
Population: Full Analysis Set - Participants with Observed Data
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cinacalcet
Number analyzed (Participants) | 161
mmol/L | -0.32 (0.02)

22. Primary Outcome: Change From Baseline to Month 6 in Albumin-corrected Serum Calcium
Time Frame: Baseline to Month 6
Population: Full Analysis Set - Participants with Observed Data
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cinacalcet
Number analyzed (Participants) | 127
mmol/L | -0.35 (0.03)

23. Primary Outcome: Change From Baseline to Month 12 in Albumin-corrected Serum Calcium
Time Frame: Baseline to Month 12
Population: Full Analysis Set - Participants with Observed Data
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cinacalcet
Number analyzed (Participants) | 109
mmol/L | -0.36 (0.03)

24. Primary Outcome: Percent Change From Baseline to Month 12 in Bone Mineral Density (g/cm^2). Anatomic Site: Femoral Neck; Densitometer: Hologic
Description: Results only shown where >10 patients have data
Time Frame: Baseline to Month 12
Population: Full Analysis Set - Participants with Observed Data
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 14
Percent change | 0.82 (5.26) [-1.63 to 2.91]

25. Primary Outcome: Percent Change From Baseline to Month 12 in Bone Mineral Density (g/cm^2). Anatomic Site: Lumbar Spine; Densitometer: Hologic
Description: Results only shown where >10 patients have data
Time Frame: Baseline to Month 12
Population: Full Analysis Set - Participants with Observed Data
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Cinacalcet
Number analyzed (Participants) | 19
Percent change | -1.16 (9.56) [-3.89 to 2.70]

26. Primary Outcome: Reason for Prescribing Cinacalcet
Time Frame: Initiation
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 303
Participants
  Failed surgery | 33 (0.9) [49.2 to 57.0]
  Surgery contraindicated | 33
  Surgery not considered appropriate by physician | 107
  Reduction of hypercalcaemia before surgery | 43
  Surgery declined by patient | 86
  Other | 1

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  Only adverse drug reactions to cinacalcet were collected. Analysis is based on the Full Analysis Set (all enrolled who fulfilled study inclusion/exclusion criteria).
Arm/Group | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 2/303
Other Adverse Events (participants affected / at risk) | 41/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=303)
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Circulatory collapse (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=303)
Nausea (Gastrointestinal disorders) | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.